CLINICAL TRIAL: NCT07305064
Title: Development and Evaluation of a Virtual Peer Agent for Psychological Counseling of Adolescents With Stressful Life Events : A Feasibility Study
Brief Title: A Virtual Peer Agent for Counseling Adolescents With Stressful Life Events
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIPeer Agent
Record Dates: First submitted 2025-11-29; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Adolescent - Emotional Problem; Agent; Psychological; Conversational
Keywords: adolescent; Stressful Life Events; Conversational agent; psychological; peer; mental health; depression
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Peer Agent Counseling (Experimental): This is the single, experimental arm of the study. All enrolled participants receive the experimental intervention, which is the virtual peer agent counseling program. This group is designed to evaluate the feasibility and preliminary efficacy of the agent-delivered support system in a real-world context, with participants completing all outcome assessments pre- and post-intervention for within-subject comparison.
  Interventions: Behavioral: Virtual Peer Agent Counseling

INTERVENTIONS:
Behavioral: Virtual Peer Agent Counseling — A conversational virtual agent designed to provide psychological support to adolescents through multi-turn dialogues. Intervention components include: psychoeducation, emotion recognition training, coping strategy development, social support exploration, and personalized behavioral task ("to-do list") setting. The intervention lasts for 4 weeks, involving multiple structured session nodes and follow-up reminders during inter-session intervals.
  Other Names: Conversational agent

SUMMARY:
This study aims to develop and evaluate a virtual companion agent for providing psychological support to adolescents who have recently experienced stressful life events. This is a single-arm, pre-post pilot trial. We plan to recruit 35 adolescents aged 14-25 to receive a 4-week intervention via the virtual agent. The intervention primarily consists of multi-turn conversations focused on helping adolescents cope with stressful events, identify emotions, enhance social support, and adopt positive coping strategies. The primary objectives are to evaluate the effectiveness of the virtual agent in improving psychological symptoms, resilience, emotional intelligence, and perceived stress, and to comprehensively assess its feasibility, acceptability, and safety.

DETAILED DESCRIPTION:
Over the past decade, mental health issues among adolescents have become increasingly prevalent. Approximately 14% of adolescents globally suffer from conditions like depression and anxiety. Adolescence is a critical developmental period, and mental health problems during this stage can have long-term negative impacts on relationships, academic performance, and future careers. However, due to factors such as cost, accessibility, and social stigma, many adolescents struggle to access timely and effective professional psychological services. In recent years, AI-based conversational agents have emerged as a potential solution. For some sensitive adolescents who are reluctant to confide in others or resistant to professional counseling, an anonymous, non-judgmental virtual conversational partner may serve as a lower-threshold avenue for them to open up and seek emotional support. Against this backdrop, this study aims to develop and evaluate a virtual companion agent specifically designed for adolescents. A minimum of 35 participants are required to complete all study procedures. Accounting for an estimated attrition rate of 20%, a total of 50 eligible adolescent participants will be enrolled. Participants will engage in a series of structured conversational interactions with the agent over 4 weeks and undergo multiple psychological assessments before, during, and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 14 and 25 years. Self-report of experiencing a stressful life event of moderate or greater severity within the past 6 months.

Total score on the relevant stress subscale of the Brief Symptom Inventory-53 (BSI-53) used for screening is < 63.

Able to understand and provide informed consent (for minor participants, informed assent from the participant and informed consent from a parent or guardian are required).

Exclusion Criteria:

* Current or previous diagnosis of a severe mental disorder (e.g., major depressive disorder, schizophrenia, bipolar disorder).

Having received more than 4 sessions of continuous professional psychotherapy or psychotropic medication treatment within the past 12 months.

Presence of severe suicidal or self-injurious behavior that is not effectively controlled and requires immediate clinical intervention.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Level of Psychological Symptoms | Baseline [week 0], Week 1 of intervention, Week 2 of intervention, Week 3 of intervention, Week 4 of intervention
  Level of Psychological Symptoms: Assessed by change in scores on the Brief Symptom Inventory-53 (BSI-53). This 53-item instrument, which encompasses 9 dimensions, is rated on a 5-point Likert scale. A cut-off point of 63 or higher is used to define a positive case.

SECONDARY OUTCOMES:
Psychological Resilience | Baseline [week 0], Week 1 of intervention, Week 2 of intervention, Week 3 of intervention, Week 4 of intervention
  Psychological Resilience: Assessed by change in scores on the Connor-Davidson Resilience Scale (CD-RISC). The instrument consists of 25 items distributed among three dimensions: Hardiness (13 items), Strength (8 items), and Optimism (4 items). Responses are recorded on a 5-point Likert scale, yielding a total score between 0 and 100, where a higher score denotes a higher level of psychological resilience.
Social Support | Baseline [week 0], Week 1 of intervention, Week 2 of intervention, Week 3 of intervention, Week 4 of intervention
  1. Social Support: Assessed by scores on the Perceived Social Support Scale (PSSS) .The Perceived Social Support Scale (PSSS) consists of 12 items, which are divided into three dimensions: family, friend, and other support. Using a 7-point Likert scale, the total score (range: 12-84) is calculated, with a higher score reflecting a higher level of perceived social support.
Emotional Intelligence | Baseline [week 0], Week 1 of intervention, Week 2 of intervention, Week 3 of intervention, Week 4 of intervention
  Description: Emotional Intelligence: Assessed by change in scores on the Wong and Law Emotional Intelligence Scale (WLEIS). The Emotional Intelligence Scale contains 16 items across four subscales: Self-Emotion Appraisal and Expression, Others' Emotion Appraisal, Regulation of Self-Emotion, and Use of Emotion. 7-point scoring system is used, and the total score for each subscale is used to determine the competency level in that specific dimension.
Coping Strategies | Baseline [week 0], Week 1 of intervention, Week 2 of intervention, Week 3 of intervention, Week 4 of intervention
  Coping Strategies: Assessed by scores on the Coping Strategy Indicator - Short Form in Chinese (CSIS-SFC).The scale is composed of 21 items divided into four subscales: Task-Oriented Coping, Emotion-Oriented Coping, Distraction Coping, and Social Diversion Coping. It is a 5-point Likert scale.
Participant Satisfaction | Within 1 week after intervention completion
  Acceptability of the virtual peer agent will be assessed using a Client Satisfaction Questionnaire (CSQ).
Session Completion Rate | Week 1 of intervention, Week 2 of intervention, Week 3 of intervention, Week 4 of intervention
  The duration of each participant's conversation per session, the total weekly interaction time, and the overall interaction time throughout the intervention period will be recorded.
Dropout Rate | From enrollment through the post-intervention assessment (at Week 4)
  Feasibility will be assessed by the study dropout rate, calculated as the percentage of participants who discontinue the study before the post-intervention assessment
User Experience | Within 1 week after intervention completion
  The overall user experience during interaction with the virtual agent will be assessed using the User Experience Questionnaire (UEQ).
Working Alliance | Within 1 week after intervention completion
  The quality of the therapeutic relationship between the participant and the virtual agent will be assessed using the Working Alliance Questionnaire(WAQ).The instrument consists of 12 items comprising three subscales: Task Goal, Emotional Bond, and Engagement. Each subscale contains 4 items and is rated on a 5-point scale.
Perceived Warmth and Professionalism | Within 1 week after intervention completion
  Participant perceptions of the virtual agent's interpersonal qualities will be assessed using scales measuring Perceived Warmth and Professionalism.

OTHER OUTCOMES:
Expert Evaluation Questionnaire | Within 1 week after intervention completion
  Safety will be assessed by an Expert Evaluation Questionnaire, where psychology experts rate the system's logic and the quality of its responses to ensure they are safe and appropriate.
High-risk Identification Match Rate | Within 1 week after intervention completion
  Safety will be assessed by the high-risk identification match rate, which measures the consistency between the virtual agent and human experts in flagging high-risk dialogue content.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request and after approval of a research proposal, de-identified individual participant data that underlie the results of this study (specifically, the pre- and post-intervention scale scores) will be made available. This does not include any raw transcript data from conversations with the virtual agent, to protect participant privacy.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After the publication of the study
Access Criteria: The researchers can access the data by contacting the PI at xiaw23@mail.sysu.edu.cn with the research purpose described.